CLINICAL TRIAL: NCT01701947
Title: HEMOLEVEN® Expanded Access Program for Prevention of Surgical and Postpartum Hemorrhage in Patients With Severe Inherited Factor XI Deficiency
Brief Title: HEMOLEVEN® Expanded Access Program Prevention of Surgical/Postpartum Hemorrhage Severe Inherited Factor XI Deficiency
Acronym: EAP
Status: No longer available | Type: Expanded Access
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: HM11-1102
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Wound; Rupture, Surgery, Cesarean Section; Postpartum Hemorrhage; Surgery
Keywords: Factor XI deficiency; EAP; postpartum hemorrhage; surgery; delivery; Child birth
MeSH Terms: conditions — Wounds and Injuries; Rupture; Postpartum Hemorrhage; Factor XI Deficiency

INTERVENTIONS:
Biological: Hemoleven — Replacement therapy
  Other Names: Human Coagulation Factor XI

SUMMARY:
The objective of the Expanded Access Program is to provide HEMOLEVEN, a replacement coagulation factor XI, to patients with severe inherited factor XI deficiency where, in the opinion of the treating physician, the benefits of administering selectively the missing factor outweigh the potential risks associated with the administration of fresh-frozen plasma.

DETAILED DESCRIPTION:
Many patients are asymptomatic until hemostatically challenged by surgery or trauma; so, the diagnosis is often made in late childhood or early adulthood but always after full liver maturation (i.e. 6 months) as reported by Andrew et al.

Spontaneous bleeding is rare, except menorrhagia, and bleeding occurs mainly after surgery or injury. Bleeding is observed mainly in surgical sites with high fibrinolytic activity such as mouth, nose, or the genitourinary tract.

Pregnancy, labor and delivery can also be challenging for women with FXI deficiency. In 1999 a study published in the American Journal of Hematology revealed that FXI levels are inconsistent during pregnancy. The incidence of postpartum hemorrhage is increased in women with factor XI deficiency. The incidence is 16% for the primary postpartum hemorrhage in FXI patients, compared with 5% in the general population. Moreover, the incidence is 24% for the secondary postpartum hemorrhage in comparison with that in the general obstetric population (0.7%). The authors recommend that FXI levels be obtained during the initial visit and monitored during the woman's third trimester. For all of these reasons it is important for women who suspect they might have a FXI deficiency to be tested and diagnosed before pregnancy.

Severe factor XI deficiency is defined by levels of <0.20 IU/mL. Such individuals have a high probability of post-operative hemorrhage. Individuals with levels between 0.20 IU/mL and the lower limit of the normal range, generally 0.65-0.80 IU/mL, are generally classified as having partial or mild deficiency with a lower risk of post-operative bleeding. Partial deficiency is being increasingly recognized following pre-operative tests or as a result of family screening. Thus partial factor XI deficiency is often diagnosed in asymptomatic individuals, creating management dilemmas because of the unpredictability of the bleeding risk. To differentiate an isolated or combined bleeding disorder in a patient with factor XI deficiency, other causes of bleeding should be investigated and excluded (e.g. von Willebrand disease, platelet disorders).

ELIGIBILITY:
Inclusion Criteria:

1. Severe inherited factor XI deficiency (FXI:C < 0.20 IU/mL i.e. <20 %)
2. Patient older than 6 months old and weight at least 8 kg
3. Known personal bleeding history
4. Patient requiring FXI replacement therapy when oral antifibrinolytic agents alone or other means are ineffective or are contraindicated
5. Scheduled to undergo an elective surgical procedure (including caesarean section) for which the patient requires hemostasis prophylaxis, which in the case of caesarean section is due to a history of postpartum bleeding, OR vaginal delivery for which the patient requires hemostasis prophylaxis due to a history of postpartum hemorrhage
6. Patient/guardian provides signed and dated Informed Consent for 'HEMOLEVEN Expanded Access Program' prior to entry into the program

Exclusion Criteria:

1. Personal history of thromboembolic events
2. Underlying cardiopulmonary disease of NYHA Class III or greater
3. History of severe reaction to any component of HEMOLEVEN notably to heparin or to its derivatives,including LMWH. Past history of serious type II heparin-induced thrombocytopenia (HIT)
4. Presence of antibody to FXI in the past or currently
5. Presence of any other condition that could contraindicate treatment with factor XI concentrate or lead the Physician/Investigator to believe treatment would not be in the best interest of the patient
6. Positive, confirmed pregnancy test for patients undergoing elective surgery (not applicable for caesarean section and prevention in vaginal delivery)
7. Lactating woman.

Of the seven exclusion criteria, the first four are included as a precautionary safety measure; the fifth is included to avoid a lack of efficacy.

The two last criteria are included to minimize confounding influences on the evaluation of patient safety. Oral contraception is not mandatory as a pregnancy test is scheduled at inclusion visit and before surgery.

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Anne T Neff, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center - Hemostasis & Thrombosis Ctr, Nashville, Tennessee, United States